CLINICAL TRIAL: NCT04798638
Title: Studies to Compare the Pharmacokinetics of TY-9591 Tablets and Osimertinib Mesylate Tablets After a Single Fasting Administration and Determine the Effect of Food on the Pharmacokinetics of TY-9591 Tablets in Healthy Volunteers
Brief Title: A Study to Assess the Effect of Food on the Pharmacokinetics of TY-9591 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TYK Medicines, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TYKM1601102
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2021-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1: TY-9591 + Osimertinib + TY-9591 (Experimental): Participants will receive TY-9591 tablets under fasted condition in period 1 , followed by Osimeritinib Mesylate tablet under fasted condition in period 2. In period 3, participants will receive TY-9591 tablet in fed state (high-fat meal). The washout will be no less than 21 days between each treatment.
  Interventions: Drug: TY-9591 Tablets under Fasted Condition - Arm1; Drug: Osimertinib Mesylate Tablets under Fasted Condition - Arm1; Drug: TY-9591 Tablets after a High-fat Meal - Arm1
- Arm2: Osimertinib + TY-9591 + TY-9591 (Experimental): Participants will receive Osimeritinib Mesylate tablet under fasted condition in period 1 , followed by TY-9591 tablets under fasted condition in period 2. In period 3, participants will receive TY-9591 tablet in fed state (high-fat meal). The washout will be no less than 21 days between each treatment.
  Interventions: Drug: Osimertinib Mesylate Tablets under Fasted Condition - Arm2; Drug: TY-9591 Tablets under Fasted Condition - Arm2; Drug: TY-9591 Tablets after a High-fat Meal - Arm2

INTERVENTIONS:
Drug: TY-9591 Tablets under Fasted Condition - Arm1 — Phase 1 (period 1) fasted from 10 hours prior to dosing with 80 mg TY-9591 tablet (p o, once) and 4 hours after dosing on day 1.
  Other Names: TY-9591
  Arms: Arm1: TY-9591 + Osimertinib + TY-9591
Drug: Osimertinib Mesylate Tablets under Fasted Condition - Arm1 — Phase 1 (period 2) fasted from 10 hours prior to dosing with 80 mg Osimertinib Mesylate Tablets (p o, once) and 4 hours after dosing on day 1.
  Other Names: AZD9291
  Arms: Arm1: TY-9591 + Osimertinib + TY-9591
Drug: TY-9591 Tablets after a High-fat Meal - Arm1 — Phase 2 (period 3) allocated high-fat meal prior to dosing with 80 mg TY-9591 tablet (p o, once) and 4 hours after dosing on day 1.
  Other Names: TY-9591
  Arms: Arm1: TY-9591 + Osimertinib + TY-9591
Drug: Osimertinib Mesylate Tablets under Fasted Condition - Arm2 — Phase 1 (period 1) fasted from 10 hours prior to dosing with 80 mg Osimertinib Mesylate Tablets (p o, once) and 4 hours after dosing on day 1.
  Other Names: AZD9291
  Arms: Arm2: Osimertinib + TY-9591 + TY-9591
Drug: TY-9591 Tablets under Fasted Condition - Arm2 — Phase 1 (period 2) fasted from 10 hours prior to dosing with 80 mg TY-9591 tablet (p o, once) and 4 hours after dosing on day 1.
  Other Names: TY-9591
  Arms: Arm2: Osimertinib + TY-9591 + TY-9591
Drug: TY-9591 Tablets after a High-fat Meal - Arm2 — Phase 2 (period 3) allocated high-fat meal prior to dosing with 80 mg TY-9591 tablet (p o, once) and 4 hours after dosing on day 1.
  Other Names: TY-9591
  Arms: Arm2: Osimertinib + TY-9591 + TY-9591

SUMMARY:
To assess the pharmacokinetics of TY-9591 tablets and Osimertinib Mesylate tablets after a single fasting administration and the effect of food on the pharmacokinetics of TY-9591 tablets in healthy volunteers.

DETAILED DESCRIPTION:
This is a single center, randomized, open label, two phases study in healthy adult volunteers. The first phase is a two-sequence, two-period crossover trial. The volunteers will be randomly distributed into two groups and given either TY-9591 tablets or Osimertinib Mesylate tablets on a single fasting administration. In the second phase, all volunteers will be administrated TY-9591 tablets after a high fat meal. The washout between each treatment is no less than 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male must be ≥ 18 and ≤ 55 years of age.
2. Bodyweight of male must be ≥ 50.0 kg (bodyweight of female must be ≥ 45.0 kg), and the Body Mass Index must be ≥ 19.0 and ≤26.0 kg/m2.
3. The participants must have no birthing plan and agree to take adequate non-drug contraceptive measures within 2 weeks before screening to 6 months after the last drug treatment.
4. The participants have good communications with investigators, understand and comply with all requirements and fully understand and sign the informed consent form.
5. The results of physical examination, vital signs, ECG, laboratory examination and other relevant examination should compliance with the clinical protocol, or they will be recognized as non-clinical signs (NCS) if beyond the regulated range.

Exclusion Criteria:

1. The participants who smoked daily >5 sticks of cigarette 3 months prior to screening or cannot give up smoking during study.
2. The participants consumed more than 14 units of alcohol per week (1 unit = 360 ml beers/45 ml liquor containing 40% alcohol/150 ml grape wine) 3 months prior to screening period, positive results of alcohol breath test and the volunteers who cannot give up drinking during study.
3. The participants who have overconsumption of tea, coffee, and the drink with caffeine (> 8 cup one day, 1 cup=250 ml) daily 3 months prior to screening period.
4. The participants have history of substance abuse and drug use within 6 months before screening.
5. The participants have history of chronic disease and serious illness in nervous system, vascular system, blood and lymphatic system, immune system, urinary system, respiratory system, digestive system and other metabolic system, any conditions and illness threat to the health of participants, and the history of hereditary disease.
6. The participants had a clinically significant disease, major surgery within 3 months before screening or plan surgery during the study period, and the surgery could affect drug absorption, distribution, metabolism, and excretion.
7. The participants who participated other clinical trials and took the investigational drug 3 months prior to first dose.
8. The participants who have blood donation or excessive bleeding (≥ 400 ml) 3 months prior to first dose, and planned to donate blood or receive blood transfusions.
9. The participants who were taking any prescription medicine, any over-the-counter (OTC), traditional chinese medicine and health care products within 14 days prior to screening period; CYP3A4 inducers/inhibitors within 30 days prior to screening period.
10. The participants who have eaten grapefruit, orange, mango, pitaya, chocolate, any caffeinated food or drink that affects the absorption, distribution, metabolism and excretion of the drug within 7 days before first dose.
11. The participants who cannot comply with the roles of unified diet.
12. The participants who have positive test result in HBsAg, antibodies against HCV (anti-HCV), Anti-HCV, Anti-HIV and TPPA.
13. The participants who cannot tolerate blood collection through venipuncture.
14. Any factors judged by investigator that the participants cannot meet.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Cmax of TY-9591 and its metabolites | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of TY-9591 and its metabolites (TY-9591-D1 (AZ5104) and TY-9591-D2) by assessment of the maximum plasma concentration.
Cmax of Osimertinib and its metabolites | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of Osimertinib and its metabolites (AZ5104 and AZ7550) by assessment of the maximum plasma concentration.
AUC(0-72h) of TY-9591 and its metabolites | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of TY-9591 and its metabolites (TY-9591-D1 (AZ5104) and TY-9591-D2) by assessment of area under the plasma concentration time curve from zero to 72 hours.
AUC(0-72h) of Osimertinib and its metabolites | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of Osimertinib and its metabolites (AZ5104 and AZ7550) by assessment of area under the plasma concentration time curve from zero to 72 hours.

SECONDARY OUTCOMES:
Tmax of TY-9591 and its metabolites | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of TY-9591 and its metabolites by assessment of time to Cmax.
Tmax of Osimertinib and its metabolites | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of Osimertinib and its metabolites by assessment of time to Cmax.
T1/2 of TY-9591 and its metabolites | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of TY-9591 and its metabolites by assessment of Terminal half life.
T1/2 of Osimertinib and its metabolites | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of Osimertinib and its metabolites by assessment of Terminal half life.
λz of TY-9591 and its metabolites | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of TY-9591 and its metabolites by assessment of Terminal rate constant.
λz of Osimertinib and its metabolites | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of Osimertinib and its metabolites by assessment of Terminal rate constant.
AUC(0-168h) of TY-9591 and its metabolites | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of TY-9591 and its metabolites by assessment of area under the plasma concentration time curve from zero to 168 hours.
AUC(0-168h) of Osimertinib and its metabolites | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of Osimertinib and its metabolites by assessment of area under the plasma concentration time curve from zero to 168 hours.
AUC(0-t) of TY-9591 and its metabolites | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of TY-9591 and its metabolites by assessment of area under the plasma concentration time curve from zero to appointed time.
AUC(0-t) of Osimertinib and its metabolites | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of Osimertinib and its metabolites by assessment of area under the plasma concentration time curve from zero to appointed time.
AUC(0-∞) of TY-9591 and its metabolites | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of TY-9591 and its metabolites by assessment of area under the plasma concentration time curve from zero to infinity.
AUC(0-∞) of Osimertinib and its metabolites | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of Osimertinib and its metabolites by assessment of area under the plasma concentration time curve from zero to infinity.
CL/F of TY-9591 | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of TY-9591 only by assessment of apparent plasma clearance.
CL/F of Osimertinib | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of Osimertinib only by assessment of apparent plasma clearance.
Vss/F of TY-9591 | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of TY-9591 only apparent volume of distribution.
Vss/F of Osimertinib | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of Osimertinib only apparent volume of distribution.
Calculated for both Cmax and AUC of TY-9591 | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of TY-9591 parent to metabolite ratio.
Calculated for both Cmax and AUC of Osimertinib | Blood samples are collected at pre-dose (within 1 hour) and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 hours post-dose.
  Pharmacokinetics of Osimertinib parent to metabolite ratio.
Safety variables | Assessments performed throughout the study period.
  Adverse events, clinical symptoms, vital signs, ECG's, clinical laboratory safety tests, ect.

CONTACTS AND LOCATIONS:
Overall Officials: Kunyan Li, Ph.D, Principal Investigator — Hunan Provincial Tumor Hospital; Xue Chen, MD, Principal Investigator — Hunan Provincial Tumor Hospital
Locations (1):
- Hunan Provincial Tumor Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No